CLINICAL TRIAL: NCT04050267
Title: Effects of Low Concentrations of Nitrous Oxide on Cognitive Functions and Reaction Time
Brief Title: Effects of Low Concentrations of Nitrous Oxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VentRes-2019-02-KR
Record Dates: First submitted 2019-05-15; First posted 2019-08-08 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Nitrous Oxide Poisoning
Keywords: nitrous oxide; tracing gas; breathing experiments; cognitive tests
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: All participants go through all study arms, in random order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control group - air (Placebo Comparator): Breathing air with 21 % of oxygen (0% nitrous oxide). Performing cognitive tests as per protocol.
  Interventions: Other: Placebo - air
- Intervention Group - 5% nitrous oxide (Experimental): Breathing 5% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide
- Intervention Group - 7% nitrous oxide (Experimental): Breathing 7% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide
- Intervention Group - 10% nitrous oxide (Experimental): Breathing 10% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide
- Intervention Group - 12% nitrous oxide (Experimental): Breathing 12% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide
- Intervention Group - 15% nitrous oxide (Experimental): Breathing 15% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide
- Intervention Group - 20% nitrous oxide (Experimental): Breathing 20% nitrous oxide in air with 21 % of oxygen. Performing cognitive tests as per protocol.
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — Breathing nitrous oxide, concentrations 5, 7, 10, 12, 15, 20 % in air with 21 % oxygen, in random order.
  Arms: Intervention Group - 10% nitrous oxide; Intervention Group - 12% nitrous oxide; Intervention Group - 15% nitrous oxide; Intervention Group - 20% nitrous oxide; Intervention Group - 5% nitrous oxide; Intervention Group - 7% nitrous oxide
Other: Placebo - air — Breathing air with 21 % oxygen, no nitrous oxide.
  Arms: Control group - air

SUMMARY:
The aim of the study is to test the effects of low concentrations of nitrous oxide on cognitive functions and reaction time in human.

DETAILED DESCRIPTION:
Nitrous oxide is a widely used gas in medicine, in standard concentrations above 50%. Its favourable physical properties and easy detectability by anaesthetic gas analysors predispose nitrous oxide to become a possible "tracing gas" for leak detection in experiments in which modified breathing system are in use. In these breathing experiments, the inspired concentrations of nitrous oxide would be well below the anaesthetic/analgesic concentrations. The aim of this study is to investigate the effects of these low concentrations of nitrous oxide (5, 7, 10, 12, 15, 20 %), compared to placebo (air, 0% nitrous oxide). The cognitive functions are tested using Digit Symbol Substitution Test, Reaction Time and Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers from the Czech Technical University

Exclusion Criteria:

* pregnancy
* allergy to nitrous oxide
* severe asthma or other severe respiratory conditions
* severe cardiovascular conditions

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Cognitive test results | Through study completion, an average of 1 year
  The results of cognitive test performed during inhalation of defined concentration of nitrous oxide. Cognitive tests: Digit Symbol Substitution Test (DSST).
Reaction Time | Through study completion, an average of 1 year
  The results of reaction time test performed during inhalation of defined concentration of nitrous oxide. Reaction Time (in seconds) using a computer-based test.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, prof., Ph.D., Study Director — Czech Technical University in Prague
Locations (1):
- Czech Technical University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No